CLINICAL TRIAL: NCT01486641
Title: Anterolateral Versus Posterolateral Approach to the Fractured Hip Arthroplasty - a Change in Approach at Sundsvall Hospital.
Brief Title: Anterolateral Versus Posterolateral Approach to the Fractured Hip Arthroplasty
Acronym: APAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sebastian-12
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2014-04

CONDITIONS: Femoral Neck Fracture
Keywords: femoral neck fracture; arthroplasty; surgical approach; anterolateral; posterolateral
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anterolateral approach (Active Comparator): Patients with a displaced femoral neck fracture operated through the anterolateral approach to the hip arthroplasty.
  Lubinus total hip arthroplasty or varikopf hemiarthroplasty.
  Interventions: Procedure: Anterolateral approach
- Posterolateral approach (No Intervention): Patients with a displaced femoral neck fracture operated through the posterolateral approach to the hip arthroplasty.
  Lubinus total hip arthroplasty or varikopf hemiarthroplasty.

INTERVENTIONS:
Procedure: Anterolateral approach — Anterolateral approach acording to Gammer for hip arthroplasty.
  Other Names: Anterolateral approach according to Gammer.; Lubinus total hip arthroplasty or varikopf hemiarthroplasty.
  Arms: Anterolateral approach

SUMMARY:
The purpose of this study is to determine whether the anterolateral in comparison to posterolateral approach to the hip arthroplasty gives an equal or better clinical results.

DETAILED DESCRIPTION:
The purpose of this study is to compare the anterolateral- to posterolateral approaches in patients suffering a displaced femoral neck fracture operated with an hip arthroplasty. Our hypothesis is that the anterolateral approach gives equal or better clinical function, health related quality of life and less complication and reoperations.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Displaced femoral neck fracture

Exclusion Criteria:

* Pathologic fracture
* Not Swedish speaker
* Not living in Västernorrlands county

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Womac | 1 year postoperatively

SECONDARY OUTCOMES:
EQ5D | 1 year postoperatively
Harris Hip Score | 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Arkan S Sayed-Noor, Principal Investigator — Umeå University
Locations (2):
- Sweden (2):
  - Sundsvall Hospital, Sundsvall, Västernorrland County
  - Department of orthopedic surgery Sundsvall Hospital, Sundsvall

IPD SHARING:
Plan to Share IPD: Yes
Publication in an international peer-review journal.
Time Frame: Publishing resultat in 2017
Access Criteria: Open Access

REFERENCES:
- [Background] Ritter MA, Harty LD, Keating ME, Faris PM, Meding JB. A clinical comparison of the anterolateral and posterolateral approaches to the hip. Clin Orthop Relat Res. 2001 Apr;(385):95-9. doi: 10.1097/00003086-200104000-00016. PMID 11302333
- [Background] Gore DR, Murray MP, Sepic SB, Gardner GM. Anterolateral compared to posterior approach in total hip arthroplasty: differences in component positioning, hip strength, and hip motion. Clin Orthop Relat Res. 1982 May;(165):180-7. PMID 7075057
- [Background] Skoldenberg O, Ekman A, Salemyr M, Boden H. Reduced dislocation rate after hip arthroplasty for femoral neck fractures when changing from posterolateral to anterolateral approach. Acta Orthop. 2010 Oct;81(5):583-7. doi: 10.3109/17453674.2010.519170. PMID 20860452